CLINICAL TRIAL: NCT03251456
Title: Tertiary Care Based Visual Developmental Diseases Management Model Among Preschool Children in China: a Cluster Randomized Controlled Trial
Brief Title: Tertiary Care for Visual Developmental Disorders in Pre-school Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yizhi Liu, Clinical Professor,director of Zhongshan Ophthalmic Center, Zhongshan Ophthalmic Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYSU-OPH-002
Record Dates: First submitted 2017-08-10; First posted 2017-08-16 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: Visual Developmental Disorders
Keywords: myopia; Tertiary Care; Pre-school Children
MeSH Terms: conditions — Myopia | interventions — Tertiary Healthcare

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tertiary care (Experimental)
  Interventions: Other: Tertiary care
- Usual care (Active Comparator)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Tertiary care — 1. Inform the parents that there are abnormalities after eye disease screening of their children, and the program of tertiary care for visual developmental disorders
  2. The children will be receiving the appropriate therapy in tertiary care and follow-up according to the clinical guidelines
  3. Six months after receiving the screening report, all the parents will be interviewed by telephone, or visiting if necessary.
  Arms: Tertiary care
Other: Usual Care — 1. Inform the parents that there are abnormalities after eye disease screening of their children
  2. Inform the parents that they should take their children to the hospital for further consultation
  3. Six months after the receiving the screening report, all the parents will be interviewed by telephone, or visiting if necessary.
  Arms: Usual care

SUMMARY:
Visual development disorders are major public health problems among children especially in China. How to find an effective and economic way to manage the larger number of children in China remains exploring. The national basic public health services of China offer visual acuity screening for preschool children for free every year. The aim of this study is to demonstrate the feasibility, cost-effective and the influence factors of compliance of tertiary care for visual developmental disorders in pre-school children after screening, and whether this disease management model is more effective and superior than the current medical care in china.

DETAILED DESCRIPTION:
Visual development disorders including amblyopia , strabismus ,refractive error are an important public health problem among children, and the visual impairment caused by visual development disorders is lifelong and can be profound. Timely discovering and treatment of visual development disorders are significant for the recovering of visual function in children. The national basic public health services of China offer the basic visual acuity screening every year for free. In this study, the investigators try to explore the cost-effective and compliance of the national basic public health services based tertiary care model for the management of visual development disorders among preschool children. This Tertiary care based on disease management model among preschool children was conducted at Yudu county, Jiangxi province, in China. Preschool vision screening relied on the national basic public health services of China (refractive errors examined by the Retinomax autorefractor). Children who failed the screening were randomized into two groups, the intervention group: their parents will be informed and transferred to an ophthalmologist and optometrist at Ophthalmic Referral Center, receiving basic eye examination and therapy (visual corrected by glasses and periodic review); The control group: their parents will be informed and suggest them to take their children to the hospital for further examination by themselves.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are aged 4-7 years and of Chinese citizen
2. Who is willing to sign the consent form
3. Children at the kindergarten will receiving the eye diseases screening of public health equalization programs in China, and there are abnormal findings after screening

Exclusion Criteria:

1. Unwilling to sign the consent form
2. Exiting eye diseases and already receiving therapies and follow up

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1114 (Actual)
Dates: Start 2017-08-18 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
The consultation rate in six month after the parents receiving the visual screening report | 6 months
  The consultation rate will be determined by the number of children who had visual screening abnormal actually go to hospital for consultation by telephone follow-up.

SECONDARY OUTCOMES:
The cost-effective of the tertiary care for visual developmental disorders | 6 months
  The cost of the disease management model will be determined by the cost per child when receiving the therapy including the travelling and medical fee, and the time they spent. And the clinical efficacy of the tertiary care for visual developmental disorders will be determined by whether or not the child receiving the appropriate therapy according to the clinical guideline.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi LIU, MD,PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University; Yangfa ZENG, MD,Master, Study Director — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Yudu, Ganzhou, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vision in Preschoolers Study Group. Preschool vision screening tests administered by nurse screeners compared with lay screeners in the vision in preschoolers study. Invest Ophthalmol Vis Sci. 2005 Aug;46(8):2639-48. doi: 10.1167/iovs.05-0141. PMID 16043831
- [Background] Hendler K, Mehravaran S, Lu X, Brown SI, Mondino BJ, Coleman AL. Refractive Errors and Amblyopia in the UCLA Preschool Vision Program; First Year Results. Am J Ophthalmol. 2016 Dec;172:80-86. doi: 10.1016/j.ajo.2016.09.010. Epub 2016 Sep 14. PMID 27640004
- [Background] US Preventive Services Task Force. Vision screening for children 1 to 5 years of age: US Preventive Services Task Force Recommendation statement. Pediatrics. 2011 Feb;127(2):340-6. doi: 10.1542/peds.2010-3177. Epub 2011 Jan 31. PMID 21282267
- [Background] Konig HH, Barry JC. Cost effectiveness of treatment for amblyopia: an analysis based on a probabilistic Markov model. Br J Ophthalmol. 2004 May;88(5):606-12. doi: 10.1136/bjo.2003.028712. PMID 15090409
- [Background] Kemper AR, Wallace DK, Patel N, Crews JE. Preschool vision testing by health providers in the United States: findings from the 2006-2007 Medical Expenditure Panel Survey. J AAPOS. 2011 Oct;15(5):480-3. doi: 10.1016/j.jaapos.2011.07.007. PMID 22108361
- [Background] Donahue SP, Arthur B, Neely DE, Arnold RW, Silbert D, Ruben JB; POS Vision Screening Committee. Guidelines for automated preschool vision screening: a 10-year, evidence-based update. J AAPOS. 2013 Feb;17(1):4-8. doi: 10.1016/j.jaapos.2012.09.012. Epub 2013 Jan 27. PMID 23360915
- [Background] Donahue SP. Prescribing spectacles in children: a pediatric ophthalmologist's approach. Optom Vis Sci. 2007 Feb;84(2):110-4. doi: 10.1097/OPX.0b013e318031b09b. PMID 17299340
- [Derived] Zeng Y, Han X, Wang D, Chen S, Zheng Y, Jiang Y, Chen X, Li Y, Jin L, Chen Q, Liang X, Zhang X, Congdon N, Liu Y. Effect of a complex intervention to improve post-vision screening referral compliance among pre-school children in China: A cluster randomized clinical trial. EClinicalMedicine. 2020 Feb 4;19:100258. doi: 10.1016/j.eclinm.2020.100258. eCollection 2020 Feb. PMID 32055790